CLINICAL TRIAL: NCT04539600
Title: Induction Chemotherapy Combined With Camrelizumab Followed by Chemoradiotherapy in Locoregionally Advanced Hypopharyngeal Cancer
Brief Title: Induction Chemotherapy Combined With Camrelizumab in Locoregionally Advanced Hypopharyngeal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhen-Wei Peng, Associate Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: hypopharyngeal SCC 002
Record Dates: First submitted 2020-09-01; First posted 2020-09-07 (Actual); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Hypopharyngeal Cancer; Immunotherapy; Induction Chemotherapy
MeSH Terms: conditions — Hypopharyngeal Neoplasms | interventions — camrelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- induction chemotherapy + anti-PD-1 antibody (Experimental): Camrelizumab (200 mg, Q3w, 2 cycles in total) combined with induction chemotherapy (taxane-containing regimen, Q3w, 2 cycles in total) followed by concurrent radiotherapy and chemotherapy.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is a type of anti-PD-1 antibody that could enhance the immune system of the patient to fight cancer.

SUMMARY:
The study is a single center phase II trial. The purpose is to investigate both the efficacy and safety of chemotherapy combined with anti-PD-1 antibody Followed by chemoradiotherapy in locoregionally advanced hypopharyngeal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years;
2. Hypopharyngeal squamous cell carcinoma confirmed by histopathology;
3. No distant metastases, stage III-IV (According to the 8th UICC/AJCC TNM staging system );
4. At least 1 measurable lesion (according to RECIST1.1), and the lesion has not been treated;
5. Provide tissues for biomarker analysis;
6. ECOG PS 0-1;
7. Adequate hematologic, hepatic and renal function: ANC ≥ 1.5x10^9/L, Hb ≥ 90g/L, PLT ≥ 100 x10^9/L, albumin ≥ 28g/L, total bilirubin < 1.5×ULN at diagnosis or after biliary drainage, ALT and AST < 5×ULN, BUN、CREA<1.5×ULN, creatinine clearance rate ≥ 45ml/min;
8. Contraception during the study;
9. At least 12 weeks of life expectancy;
10. Willing to join the study and sign informed consent.

Exclusion Criteria:

1. Allergic to any component of carrelizumab, cisplatin and other platinum drugs;
2. Have received anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137 or CTLA-4 antibody therapy in the past;
3. Received biological treatment or participated in clinical trial of other drugs or devices within 4 weeks before enrollment;
4. Have other malignant tumors within 5 years, except for fully treated basal cell/squamous cell skin cancer/cervical cancer;
5. Have corticosteroids (>10 mg prednisone equivalent dose per day) or other immunosuppressive agents for systemic treatment within 2 weeks before the first use of the study drug, except for local inflammation and prevention of allergies, nausea or vomiting;
6. Uncontrolled clinical symptoms or diseases of the heart, such as: heart failure above NYHA II, unstable angina, myocardial infarction within 1 year；
7. Have severe infections (CTCAE> Grade 2) occurred within 4 weeks before the first use of the study drug;
8. Have active autoimmune diseases, autoimmune diseases, but not including autoimmune-mediated hypothyroidism treated with stable doses of thyroid replacement hormone; type 1 diabetes with stable doses of insulin; vitiligo or cured childhood asthma/allergies;
9. A history of immunodeficiency, including a positive HIV test, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
10. A history of interstitial lung disease (excluding radiation pneumonia that has not been treated with hormones) and a history of non-infectious pneumonia;
11. Active tuberculosis, having antituberculosis therapy at present or within 1 year;
12. Have active hepatitis B (HBV DNA ≥2000 IU/mL or 10~4 copies/mL) and hepatitis C;
13. Have other uncontrollable comorbidities;
14. Knowing a history of psychotropic drug abuse, alcohol or drug abuse;
15. Pregnant or breastfeeding, or expect to become pregnant during the clinical trial period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-12-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival, PFS | 1 year
  Defined as the time from randomization until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  Defined as the portion of patients with a tumor size reduction of a predefined amount for a minimum time period. Tumor response will be measured according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1.
Duration of Response（DoR） | 1 year
  Response duration is measured from the time of initial response until documented tumor progression.
Disease Control Rate (DCR) | 1 year
  Refers to the proportion of patients whose tumors have shrunk or been stable for a certain period of time, including cases of complete response (CR), partial response (PR), or stable disease (SD).
Overall Survival (OS) | 1 year
  Defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.
Adverse events (AE) | 1 year
  Adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided